CLINICAL TRIAL: NCT01848223
Title: The Quality of Life in Late Menopause. A Seventeen Years Follow-up Study.
Brief Title: The Quality of Life in Late Menopause
Acronym: QoL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: T56/2013
Record Dates: First submitted 2013-05-02; First posted 2013-05-07 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Quality of Life
Keywords: quality of life; QoL; late menopause

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- late menopause

SUMMARY:
The purpose of this study is to evaluate the quality of life of late postmenopausal Finnish women and the factors affecting it.

DETAILED DESCRIPTION:
The aim of this study is to investigate the quality of life (QoL) of late postmenopausal Finnish women. In 1995, 71 women were recruited through an advertisement in a local newspaper in the area of Turku in Finland. Exclusion criteria were: a history of previous head injury, neurological, cardiovascular, endocrinological or mental disease, medicated hyperlipidemia, malignancies, abuse of alcohol or medicines and smoking (over 10 cigarettes daily). Inclusion criteria were: previous hysterectomy for a benign reason and postmenopausal status (serum follicle stimulating hormone (FSH) level over 26 U/l). Finally, 65 women were approved for the study.

Originally the study was a prospective, randomized, placebo-controlled, double-blind, cross-over trial. It included three different periods in which different medications were administered: three months of estrogen/placebo therapy, a one month wash-out period and three months of placebo/estrogen therapy. The women were randomized into two groups, where the other group received first a placebo and then estrogen and the other received first estrogen and then a placebo. Women completed questionnaires at the beginning of the study and after the both periods. After the survey women got to choose if they wanted to continue with the hormone replacement therapy (HRT) or not.

Questionnaires were sent to the same women six years later. The intention was to estimate the present QoL of the women. Also their use of HRT, possible chronic diseases and medications were evaluated.

This study is the 17 year follow-up study to the investigation described above. The goal is to measure the QoL of the same women and estimate the factors affecting it in late postmenopausal age. The questionnaires used are the Women's Health Questionnaire (WHQ), the Beck Depression Inventory (BDI), the Basic Nordic Sleep Questionnaire (BNSQ) and a common questionnaire to define the women's current life situation, their education and working background, their state of health, medications, the use of HRT and recent life events. The women also filled in the same questionnaires 17 years ago in relation to the first part of the study, and six years after it relating to the first follow-up study. The results of this study are compared to the former investigation results. The above mentioned randomization system is not used this time but the women are processed as only one group. The women are now acting as their own controls and their answers are compared to the responses they gave 17 years earlier. In this way it is possible to determine, if the woman's QoL has changed during aging, and if the change is for the better or worse. The women were already postmenopausal 17 years ago, so the effect of climacterium should be bypassed by now. Therefore, when the results of this study are compared to the former results, it is possible to separate the effect of the climacterium, and on the other hand, the effects of aging, on the QoL and on some symptoms attached to the perimenopausal phase.

ELIGIBILITY:
Inclusion Criteria:

* a previous hysterectomy for benign reason
* postmenopausal status (serum follicle stimulating hormone (FSH) level over 26 U/l)

Exclusion Criteria:

* a history of previous head injury
* a chronic somatic or mental disease
* abuse of alcohol or medicines
* smoking (over 10 cigarettes daily)

Ages: 64 Years to 82 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: community sample of the area of Turku
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-05 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
quality of life | seventeen years

CONTACTS AND LOCATIONS:
Overall Officials: Riina Katainen, MD, Principal Investigator — University of Turku and Turku University Hospital; Päivi Polo, MD,PhD, Study Director — University of Turku and Turku University Hospital
Locations (1):
- University of Turku and Turku University Hospital, Turku, Finland